CLINICAL TRIAL: NCT04488120
Title: A Randomized, Controlled,Multi-Centre Trial of the Efficacy and Safety of the Occlutech Septal Occluder(Figulla Flex II) Compared to the AGA Septal Occluder(Amplatzer ASO) for Transcatheter Closure of Secundum ASD in Patients
Brief Title: Occlutech Septal Occluder (Figulla Flex II) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Occlutech International AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Occ201201
Record Dates: First submitted 2020-07-20; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Secundum Atrial Septal Defects
Keywords: Occlutech; Transcatheter closure of secundum atrial septal defects; Figulla Flex II; Occ201201

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, multi-centre trial of the efficacy and safety of the Occlutech septal occluder (Figulla Flex II) compared to the AGA septal occluder (Amplatzer ASO) for transcatheter closure of secundum atrial septal defects in patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Occlutech septal occluder ( Figulla Flex II) (Experimental): Occlutech septal occluder (Figulla Flex II)
  Interventions: Device: transcatheter closure of secundum atrial septal defects in patients
- Amplatzer Septal Occluder (ASO) (Active Comparator): St. Jude AGA septal occluder (Amplatzer ASO)
  Interventions: Device: transcatheter closure of secundum atrial septal defects in patients

INTERVENTIONS:
Device: transcatheter closure of secundum atrial septal defects in patients — transcatheter closure of secundum atrial septal defects in patients

SUMMARY:
The objectives of the study are:

* To determine the efficacy of the Figulla Flex II device compared with that of the Amplatzer ASO device for transcatheter closure of secundum atrial septal defects
* To determine the safety of the Figulla Flex II device compared with that of the Amplatzer ASO device for transcatheter closure of secundum atrial septal defects

This is a randomized, controlled, multi-centre trial of the efficacy and safety of the Occlutech septal occluder (Figulla Flex II) compared to the AGA septal occluder (Amplatzer ASO) for transcatheter closure of secundum atrial septal defects in patients.

DETAILED DESCRIPTION:
Inclusion criteria A patient will be eligible for study participation if he/she meets the following criteria:

1. Able to fluently speak and understand the language in which the study is being conducted
2. Has ostium secundum atrial septal defect
3. Has a defect hole with a diameter of < 38 mm
4. Has a left-to-right shunt with a Qp/Qs ratio of . 1.5:1 or the presence of right ventricular volume overload determined by transthoracic echo (TTE) or clinical symptoms due to the atrial septal defect
5. Has a distance of > 5 mm from the margins of the defect(s) to the coronary sinus, arterioventricular (AV) valves and right upper pulmonary vein as measured by echocardiography
6. Agrees to participate in the study and comply with the follow-up schedule
7. Is willing to freely give (or Legally Authorized Representative is willing to freely give) Informed Consent prior to treatment
8. Willing to return for the post-treatment evaluation. Exclusion criteria

A patient will be excluded from the study if he/she meets the following criteria:

1. Has multiple defects which can�ft adequately be covered by the device
2. Has associated congenital cardiac anomalies which require cardiac surgery

   a. Has a known sensitivity to contrast media that cannot be controlled adequately with pre-medication.
3. Patient is currently participating in another clinical device or drug trial that has not completed its primary endpoint or that will clinically confound the current study endpoints or does not permit subjects to participate in other studies. Typically, subjects that are involved in the long-term surveillance phase of a clinical study are eligible.
4. Has ostium primum atrial septal defects
5. Has sinus venosus atrial septal defects
6. Has partial anomolous pulmonary venous drainage
7. Has pulmonary vascular resistance above 7 Woods units or a right-toleft shunt at the atrial level with a peripheral arterial saturation less than 94%
8. Has a recent myocardial infarction, unstable angina and decompensated congestive heart failure (CHF)
9. Has right and/or left ventricular decompensation with ejection fraction of < 30%
10. Has an active bacterial and/or viral infection
11. Has any type of serious infection < 1 month prior to the procedure
12. Has malignancy where life expectancy is < 2 years
13. Has demonstrated intracardiac thrombi on echocardiography
14. Weighs < 8 kg
15. Has gastritis, gastric ulcer, duodenal ulcer, etc. and other contraindications to aspirin therapy unless other anti-platelet agents can be administered for 6 months
16. Has an unstable condition or otherwise thought to be unreliable or incapable of complying with the requirements of the clinical investigational plan (CIP).
17. Has any disorder that, in the opinion of the Investigator, might interfere with the conduct of the study.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for study participation if he/she meets the following criteria:

1. Able to fluently speak and understand the language in which the study is being conducted
2. Has ostium secundum atrial septal defect
3. Has a defect hole with a diameter of < 38 mm
4. Has a left-to-right shunt with a Qp/Qs ratio of ≥ 1.5:1 or the presence of right ventricular volume overload determined by transthoracic echo (TTE) or clinical symptoms due to the atrial septal defect
5. Has a distance of > 5 mm from the margins of the defect(s) to the coronary sinus, arterioventricular (AV) valves and right upper pulmonary vein as measured by echocardiography
6. Agrees to participate in the study and comply with the follow-up schedule
7. Is willing to freely give (or Legally Authorized Representative is willing to freely give) Informed Consent prior to treatment
8. Willing to return for the post-treatment evaluation

Exclusion Criteria:

1. Has multiple defects which can't adequately be covered by the device
2. Has associated congenital cardiac anomalies which require cardiac surgery

   a. Has a known sensitivity to contrast media that cannot be controlled adequately with pre-medication.
3. Patient is currently participating in another clinical device or drug trial that has not completed its primary endpoint or that will clinically confound the current study endpoints or does not permit subjects to participate in other studies. Typically, subjects that are involved in the long-term surveillance phase of a clinical study are eligible.
4. Has ostium primum atrial septal defects
5. Has sinus venosus atrial septal defects
6. Has partial anomolous pulmonary venous drainage
7. Has pulmonary vascular resistance above 7 Woods units or a right-toleft shunt at the atrial level with a peripheral arterial saturation less than 94%
8. Has a recent myocardial infarction, unstable angina and decompensated congestive heart failure (CHF)
9. Has right and/or left ventricular decompensation with ejection fraction of < 30%
10. Has an active bacterial and/or viral infection
11. Has any type of serious infection < 1 month prior to the procedure
12. Has malignancy where life expectancy is < 2 years
13. Has demonstrated intracardiac thrombi on echocardiography
14. Weighs < 8 kg
15. Has gastritis, gastric ulcer, duodenal ulcer, etc. and other contraindications to aspirin therapy unless other anti-platelet agents can be administered for 6 months
16. Has an unstable condition or otherwise thought to be unreliable or incapable of complying with the requirements of the clinical investigational plan (CIP).
17. Has any disorder that, in the opinion of the Investigator, might interfere with the conduct of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2012-05-21 (Actual); Primary Completion 2015-12-23 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Efficacy: the rate of a successful placement of the device | the day after procedure but no later than 36 hours after the procedure.
  The primary efficacy endpoint was early efficacy success rate, which was defined as the rate of a successful placement of the device, and successful closure of the defects without major complication, surgical reintervention, device embolization or moderate or large residual shunt the day after procedure but no later than 36 hours after the procedure.
Efficacy:The secondary efficacy endpoint is the rate of closure success (residual shunt is smaller than or equal to 2 mm) within 6 months after the procedure, without the need for surgical repair. | within 6 months after the procedure
  The secondary efficacy endpoint is the rate of closure success (residual shunt is smaller than or equal to 2 mm) within 6 months after the procedure, without the need for surgical repair.
Efficacy:Other efficacy endpoint was the rate of complete closure (no residual shunt) at 6 months after the procedure. | at 6 months after the procedure.
  Other efficacy endpoint was the rate of complete closure (no residual shunt) at 6 months after the procedure.

SECONDARY OUTCOMES:
Safety: Major, minor complications rate, all SAEs | 6 and 12 months post procedure
  Major and complications rate

IPD SHARING:
Plan to Share IPD: Undecided